CLINICAL TRIAL: NCT00234312
Title: Escitalopram vs. Sertraline in the Treatment of Dysthymic Disorder and Double Depression
Brief Title: Medications for the Treatment of Dysthymic Disorder and Double Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Joshua Boverman, MD, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 04-2801-A 02
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Depression; Dysthymia
Keywords: Depressive Disorders
MeSH Terms: conditions — Depression; Dysthymic Disorder; Depressive Disorder | interventions — Escitalopram; Sertraline

INTERVENTIONS:
Drug: escitalopram and sertraline

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of flexible doses of escitalopram (Lexapro) compared to sertraline (Zoloft) for treatment of Dysthymic Disorder.

DETAILED DESCRIPTION:
Dysthymic Disorder is a common, chronic type of depression that is often seen as a mild condition and is under-treated. Because of its chronic course, it is often complicated by episodes of major depression and may require long-term treatment.

This is a twelve week study during which daily doses of escitalopram (10-20 mg) or sertraline (50-200 mg) will be given to outpatients meeting criteria for Dysthymic Disorder or Double Depression. Medications will be assigned 1:1 and clinicians will be blinded to treatment. Efficacy will be based on scores for the Hamilton Depression Rating Scale, patient subjective reporting, and clinician observation. The study will have a total of 8 visits over 12 weeks, with a one-week medication taper period at the end. Subjects will have a physical exam, labs, and vital signs monitored at first visit and vital signs monitored at every subsequent visit. Women of childbearing potential must have a negative urine pregnancy test at screening. All subjects will remain on the lowest medication dose for the first four weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Dysthymic Disorder or Major Depressive Disorder with Antecedent Dysthymia
* Women of childbearing potential must have negative pregnancy test at screen and agree to practice acceptable method of birth control
* Score of at least 12 on the 24-item Hamilton Depression Scale at study entry
* Initial screening labs grossly within normal limits
* Signed written informed consent

Exclusion Criteria:

* Other Axis-I diagnoses such as delirium, dementia, and substance dependence (active in last year) or any substance abuse including alcohol within the past six months
* Actively suicidal
* CNS neoplasm, demyelinization disease, degenerative neurological disorder, active CNS infection, or any progressive CNS disorder that may confound interpretation of study results
* History of seizure disorder, or EEG showing paroxysmal activity or head CT showing gross structural abnormality
* Acute systemic medical disorder
* Use of any psychotropic medications within 2 weeks prior to screen or 4 weeks prior to screen in the case of fluoxetine
* Current use of any herbal medication such as St. John's wort,
* Uncontrolled renal, hepatic, endocrine, cardiovascular, pulmonary, immunological, hematological or gastrointestinal disease
* Any other abnormal medical screening tests judged by the investigator to be clinically significant
* Received any experimental medication within 30 days prior to study entry
* Patients presently in or soon to be starting psychotherapy
* Prior treatment non-response to an adequate trial of citalopram, escitalopram, or sertraline
* History of allergy to citalopram, escitalopram or sertraline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-09 (Actual); Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
score on first 17 items of HAM-D Rating Scale 24 item, each visit

SECONDARY OUTCOMES:
scores on HAM-D 21, HAM-D 24, and Beck Depression Inventory (pt. rated)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Boverman, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States